CLINICAL TRIAL: NCT01011543
Title: Comparison of Induced Sputum and Bronchoscopic Approach (BAL, Fluoroscopy-guided Transbronchial Biopsies) in Patients Suspected of Pulmonary Tuberculosis With Negative Direct Exam on Three Consecutive Non-induced Sputum Samples
Brief Title: Induced Sputum Versus Bronchoscopy in Smear Negative Pulmonary Tuberculosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: B07620096009
Record Dates: First submitted 2009-10-05; First posted 2009-11-11 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2015-08

CONDITIONS: Pulmonary Tuberculosis
Keywords: pulmonary tuberculosis; negative sputum exam; induced sputum; endoscopy
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Bronchoscopy; Bronchoalveolar Lavage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endoscopic approach (Active Comparator): CT thorax is done in all patients to localize the exact anatomical site of the disease. This evaluation is followed by fluoroscopy-guided bronchoscopy for BAL (bronchoalveolar lavage) and TBB (transbronchial biopsies). A sputum sample immediately after the endoscopy will be collected if possible.
  Interventions: Procedure: Diagnostic techniques in pulmonary tuberculosis
- Induced sputum (Active Comparator): Sputum induction after administration of 6-8 mL 3% NaCl aerosol by an ultrasonic nebulizer; sputum will be collected 15-30 minutes after administration of the aerosol. This process will be done twice in every patient.
  Interventions: Procedure: Diagnostic techniques in pulmonary tuberculosis

INTERVENTIONS:
Procedure: Diagnostic techniques in pulmonary tuberculosis — Two different methods to obtain a diagnosis of pulmonary tuberculosis in patients with negative classic sputum samples are compared.
  Other Names: Bronchoscopy; Fluoroscopy-guided bronchoscopy; Bronchoalveolar lavage; Sputum induction

SUMMARY:
This is a randomised study that compares different diagnostic approaches for diagnosing pulmonary tuberculosis in patients suspected of pulmonary tuberculosis in whom the three classic (non-induced) sputum samples didn't show tuberculous bacillus on direct examination.

The investigators compare the sensibility of induced sputum technique with an endoscopic approach (CT-scan followed by BAL and fluoroscopy-guided transbronchial biopsies and eventually sputum collection immediately after the bronchoscopy).

People in high risk population for tuberculosis undergoing screening by chest X-ray or symptomatic patients will be admitted to the hospital if their chest X-ray shows a suspicion of active tuberculosis.

According good clinical practice: (non-induced) sputum samples will be taken at admission and every following morning. If direct examination and PCR of the first three classic sputum samples are negative: patients will be randomised in two groups with a different diagnostic approach (induced sputum versus endoscopic approach) The aim of our study is to proof that a thoroughgoing endoscopic approach has a higher sensibility than an induced sputum in the diagnosis of pulmonary tuberculosis in patients with a high suspicion of active tuberculosis on the chest X-ray but with a negative direct examination and/or PCR on three consecutive normal sputum samples.

The investigators will include 154 patients (based on a statistical analysis for a hypothesis that the endoscopic approach has a sensibility that's twice the sensibility of the induced sputum).

* first arm: 2 consecutive induced sputum using an ultrasonic nebulizer.
* second arm: CT thorax to evaluate the exact anatomic localisation of the disease followed by fluoroscopy-guided bronchoscopy for BAL (bronchoalveolar lavage) and transbronchial biopsies. A sputum sample immediately after the endoscopy will be collected if possible.

ELIGIBILITY:
Inclusion Criteria:

* Patient suspected of pulmonary tuberculosis with 3 consecutive (non-induced) sputum samples negative on direct exam and PCR.

Exclusion Criteria:

* Age < 18
* Pregnancy
* Actual asthma exacerbation
* Participation to study refused by patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Sensibility of diagnosis of tuberculosis (positive culture and/or PCR) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Inge M Muylle, Principal Investigator — CHU St Pierre Brussels
Locations (1):
- CHU St Pierre; pulmonology department, Brussels, Belgium